CLINICAL TRIAL: NCT02752659
Title: Reliability and Validity of Self-measured Arm Circumference in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kristin Campbell, Associate Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H16-00961
Record Dates: First submitted 2016-04-18; First posted 2016-04-27 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Lymphedema; Breast Cancer
Keywords: Monitoring
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Women with breast cancer-related lymphedema (Experimental): Participants will measure their own arm circumference and be measured by a specialized physiotherapist and by a perometer.
  Interventions: Procedure: Self-measured arm circumference, therapist-measured arm-circumference, perometer-measured arm circumference
- Women at risk of breast cancer-related lymphedema (Experimental): Participants will measure their own arm circumference and be measured by a specialized physiotherapist and by a perometer.
  Interventions: Procedure: Self-measured arm circumference, therapist-measured arm-circumference, perometer-measured arm circumference

INTERVENTIONS:
Procedure: Self-measured arm circumference, therapist-measured arm-circumference, perometer-measured arm circumference

SUMMARY:
Early detection and treatment of onset or worsening of breast cancer-related lymphedema (BCRL) can potentially prevent or postpone the condition to progress into a chronic progressive condition or eliminate the risk of infections in the arm (cellulitis). Self-surveillance for BCRL by routinely measuring own arm circumference could potentially enable early detection of onset or worsening of lymphedema. The aim is to determine whether women who have received surgery for breast cancer, can perform self-measures of arm circumference in a reliable and valid manner using written and video supported instructions without in-person teaching by a physiotherapist.

DETAILED DESCRIPTION:
Purpose: to test the reliability and validity of self-measured arm circumference compared to measures performed by a specialized therapist and by the perometer (gold standard).

The hypothesis is that there will be an excellent correlation between arm circumference measures performed by the participant and by an experienced physiotherapist and a moderate correlation between arm circumference measures performed by the patient and determined by perometer, as well as arm volume calculated from arm circumference measurements and measured by the perometer.

Design: A cross-sectional study of women at risk of breast cancer-related lymphedema (BCRL) (n=20) and with BCRL (n=20)

Procedures: Participants will complete one self-assessment at home and one self-assessment at a laboratory the University of British Columbia (UBC).

Home Self-assessment: Participants will be sent a study package by mail, which will contain the consent form, a tape measure, written instructions supplemented with illustrations, a link for a video guide, and a measurement form, along with an opaque envelop for the measurement form. Participants will be asked to first review the written and video material outlining the measurement process, prior to completing a short self-assessment quiz on the self-measurement technique. Participants will then perform arm circumference measures of both arms as per the instructions, record the measurements on the provided form and seal the form in a provided envelope. The envelope will be returned to the study team at the lab assessment.

Lab Self-assessment: At the visit at UBC, participants will be asked by study staff to repeat these arm circumference measures with support from the video and written instructions, unsupervised by a physiotherapist. This will be followed by an assessment by the physiotherapist and measures with the perometer.

Statistical analysis plan: Intra-rater (between self-measures performed at home and at the lab), inter-rater reliability (between self-measures performed at lab and therapist-measures) and concurrent validity analysis (between self-measures performed at lab and perometer measures) will be conducted separately for women with and without BCRL.

ELIGIBILITY:
Inclusion Criteria:

* women, who have received surgery for breast cancer with axillary or sentinel lymph node dissection within the last 3 months to 5 years, including those who are undergoing chemotherapy or radiation
* with and without a clinical diagnosis of BCRL in one or two arms
* age 18 to 80 years
* who can understand the self-measurement instructions given in English
* who have access and ability to use internet to view the self-measurement video tutorial

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Intra-class correlation coefficients (ICC) for intra-rater reliability of self-measured arm circumference | Self-measures performed twice with 2 days apart
  ICC is scored from 0 to 1. Reliability is considered poor when the ICC < 0.40, moderate between 0.40 and 0.75, substantial between 0.75 and 0.90, and excellent when >0.90. The total agreement between self-measured arm circumference performed twice by the participant will be calculated.
Intra-class correlation coefficients (ICC) for inter-rater reliability between arm circumference measures performed by the participant herself and by the therapist. | Both measures are performed same day within one hour
  The total agreement between self-measured arm circumference performed by the participant and by a physiotherapist will be calculated.
Intra-class correlation coefficients (ICC) for concurrent validity of self-measured arm circumference and perometer-measures | Both measures are performed same day within one hour
  The total agreement between self-measured arm circumference performed by the participant and by a perometer will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Rafn BS, McNeely ML, Camp PG, Midtgaard J, Campbell KL. Self-Measured Arm Circumference in Women With Breast Cancer Is Reliable and Valid. Phys Ther. 2019 Feb 1;99(2):240-253. doi: 10.1093/ptj/pzy117. PMID 30289500